CLINICAL TRIAL: NCT01866163
Title: LEO 90100 Compared to Vehicle in Subjects With Psoriasis Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LP0053-1001
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Results first posted 2016-05-09 (Estimated); Last update posted 2025-03-10 (Actual); Status verified 2019-09

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LEO 90100 (Experimental): LEO 90100 aerosol foam, containing calcipotriol 50 mcg/g plus betamethasone 0.5 mg/g (as dipropionate)
  Interventions: Drug: LEO 90100
- Vehicle (Placebo Comparator): Aerosol foam vehicle
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: LEO 90100
  Arms: LEO 90100
Drug: Vehicle
  Arms: Vehicle

SUMMARY:
The purpose of this trial is to compare the efficacy of treatment with LEO 90100 to that of treatment with vehicle for up to 4 weeks in subjects with psoriasis vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of psoriasis vulgaris of at least 6 months duration involving the trunk and/or limbs
* Psoriasis vulgaris on the trunk and/or limbs (excluding psoriasis on the genitals and skin folds) involving 2-30% of the Body Surface Area (BSA)
* An Investigator's Global Assessment of disease severity (IGA) of at least mild at Day 0 (Visit 1)
* A modified PASI (m-PASI) score of at least 2 at Day 0 (Visit 1)
* A target lesion of a minimum of 5 cm at its longest axis and preferably not located on the extensor surface on an elbow or knee, scoring at least 1 for each of redness, thickness and scaliness, and at least 4 in total by the Investigator's Assessment of Severity of the Target Lesion

Exclusion Criteria:

* Systemic treatment with biological therapies, whether marketed or not, with a possible effect on psoriasis vulgaris within the following time periods prior to randomisation:

  * etanercept - within 4 weeks prior to randomisation
  * adalimumab, infliximab - within 8 weeks prior to randomisation
  * ustekinumab - within 16 weeks prior to randomisation
  * other products - within 4 weeks/5 half-lives prior to randomisation (whichever is longer)
* Systemic treatment with all other therapies with a possible effect on psoriasis vulgaris (e.g., corticosteroids, retinoids, methotrexate, ciclosporin and other immunosuppressants) within 4 weeks prior to randomisation.
* Subjects who have received treatment with any nonmarketed drug substance (i.e. a drug which has not yet been made available for clinical use following registration) within 4 weeks/5 half-lives (whichever is longer) prior to randomisation.
* PUVA therapy within 4 weeks prior to randomisation.
* UVB therapy within 2 weeks prior to randomisation.
* Topical anti-psoriatic treatment on the trunk and limbs (except for emollients) within 2 weeks prior to randomisation.
* Topical treatment on the face, scalp and skin folds with corticosteroids, vitamin D analogues or prescription shampoos within 2 weeks prior to randomisation.
* Planned initiation of, or changes to, concomitant medication that could affect psoriasis vulgaris (e.g. beta blockers, antimalarial drugs, lithium, ACE inhibitors) during the trial.
* Current diagnosis of guttate, erythrodermic, exfoliative or pustular psoriasis.
* Previously randomised in this trial or any previously conducted trial of LEO 90100.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2013-06; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Leonardi, Principal Investigator — Central Dermatology
Locations (1):
- Central Dermatology, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Veverka KA, Hansen JB, Yaloumis M, Kircik L, Stein Gold L. Calcipotriene Plus Betamethasone Dipropionate Foam for Mild Psoriasis: Pooled Results from Three Randomized Trials. J Drugs Dermatol. 2021 Aug 1;20(8):822-828. doi: 10.36849/JDD.5743. PMID 34397196
- [Derived] Iversen L, Kurvits M, Snel-Prento AM, Menter A. Calcipotriol/Betamethasone Dipropionate Cutaneous Foam Treatment for Psoriasis in Patients With BSA 5-15% and PGA >/= 3: Post-Hoc Analysis From Three Randomized Controlled Trials. Dermatol Ther (Heidelb). 2020 Oct;10(5):1111-1120. doi: 10.1007/s13555-020-00419-2. Epub 2020 Aug 12. PMID 32785881
- [Derived] Stein Gold L, Villumsen J, Rosen M. Calcipotriol Plus Betamethasone Dipropionate Aerosol Foam is Effective, Independent of Body Mass Index and the Extent and Severity of Psoriasis. Dermatol Ther (Heidelb). 2016 Dec;6(4):667-673. doi: 10.1007/s13555-016-0147-0. Epub 2016 Oct 6. PMID 27714595
- [Derived] Leonardi C, Bagel J, Yamauchi P, Pariser D, Xu Z, Olesen M, Osterdal ML, Stein Gold L. Efficacy and Safety of Calcipotriene Plus Betamethasone Dipropionate Aerosol Foam in Patients With Psoriasis Vulgaris--a Randomized Phase III Study (PSO-FAST). J Drugs Dermatol. 2015 Dec;14(12):1468-77. PMID 26659941
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Subject First Visit: 17-Jun-2013 Last Subject Last Visit: 02-Oct-2013
Pre-assignment Details: Prior to randomisation, the subject entered a washout phase (if required) where anti-psoriatic treatment and other relevant medication/treatments were discontinued as defined by the exclusion criteria. The wash-out/screening phase could last for up to 4 weeks, depending on which disallowed treatments the subject received.
Period: Overall Study
Arm/Group | LEO 90100 | Vehicle
Started | 323 | 103
Completed | 313 | 99
Not Completed | 10 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LEO 90100 | Vehicle | Total
Number analyzed (Participants) | 323 | 103 | 426
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (13.9) | 46.0 (13.2) | 50.0 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 54 | 173
  Male | 204 | 49 | 253

OUTCOME MEASURES:

1. Primary Outcome: Treatment Success According to IGA
Description: Subjects with 'treatment success' ('clear' or 'almost clear' for subjects with at least moderate disease at baseline, 'clear' for subjects with mild disease at baseline) according to the Investigators' global assessment of disease severity (IGA) at Week 4.
  The 5 point IGA scale: 1 = clear, 2 = almost clear, 3 = mild, 4 = moderate and 5 = severe
Time Frame: 4 weeks
Population: All randomised subjects were included in the full analysis set and analysed for efficacy.
Measure: Number; unit: percentage of subjects
Arm/Group | LEO 90100 | Vehicle
Number analyzed (Participants) | 323 | 103
percentage of subjects | 53.3 | 4.8
Statistical Analysis 1: Comparison: LEO 90100 vs Vehicle; Multiple imputations were used to handle missing data; Test type: Superiority or Other; p < 0.001, Mantel Haenszel; Odds Ratio (OR) = 30.27, 95% CI 2-sided [9.72 to 94.30]

2. Secondary Outcome: m-PASI at Week 4
Description: The investigator assessed the extent and severity of the three clinical signs (redness, thickness, and scaliness) on the arms, trunk and legs. These assessments were converted to an Modified Psoriasis Area and Severity Index (m-PASI).
  m-PASI (excluding head) assessed at week 4 (adjusted for the effect of (pooled) centre and baseline m-PASI.
  The m-PASI score range from 0 (best) to 64.8 (worst).
Time Frame: 4 weeks
Population: All randomised subjects were included in the full analysis set and analysed for efficacy.
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | LEO 90100 | Vehicle
Number analyzed (Participants) | 323 | 103
Scores on a scale | 2.04 [1.74 to 2.35] | 5.33 [4.79 to 5.86]
Statistical Analysis 1: Comparison: LEO 90100 vs Vehicle; The mean value and CIs were adjusted for the effect of pooled centres and baseline m-PASI. Multiple imputation was used to handle missing data; Test type: Superiority or Other; p < 0.001, ANOVA; Mean Difference (Final Values) = -3.28, 95% CI 2-sided [-3.90 to -2.67]

3. Secondary Outcome: m-PASI at Week 1
Description: as for outcome 2
Time Frame: 1 week
Population: All randomised subjects were included in the full analysis set and analysed for efficacy.
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | LEO 90100 | Vehicle
Number analyzed (Participants) | 323 | 103
Scores on a scale | 4.66 [4.41 to 4.90] | 5.93 [5.50 to 6.36]
Statistical Analysis 1: Comparison: LEO 90100 vs Vehicle; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA; Mean Difference (Final Values) = -1.27, 95% CI 2-sided [-1.76 to -0.78]

ADVERSE EVENTS:
Arm/Group | LEO 90100 | Vehicle
Serious Adverse Events (participants affected / at risk) | 2/323 | 0/103
Other Adverse Events (participants affected / at risk) | 18/323 | 15/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEO 90100 (N=323) | Vehicle (N=103)
Substance induced psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.6% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEO 90100 (N=323) | Vehicle (N=103)
Nasopharyngitis (Infections and infestations) | 6 (6) | 0 (0)
Application site pain (General disorders) | 3 (4) | 2 (2) — General disorders and administration site conditions
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Blood pressure increased (Investigations) | 3 (4) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Application site dryness (General disorders) | 0 (0) | 1 (1)
Application site erosion (General disorders) | 0 (0) | 1 (1)
Application site erythema (General disorders) | 0 (0) | 1 (1)
Application site oedema (General disorders) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO acknowledges the investigators' right to publish the results of the trial, irrespective of outcome. Pubs/presentations by investigator(s) shall not be made before the results of a joint publication is public. LEO retains the right to have any publication submitted to LEO for review. Investigators must undertake not to submit any part of their individual data for publication without the prior consent of LEO.